CLINICAL TRIAL: NCT07380867
Title: Localization of Preoperative Endoscopic Tattooing Using Indocyanine Green(ICG)-Hyaluronic Acid Mixture (Luminomark) for Colorectal Cancer Surgery
Brief Title: Confirming the Accuracy of Endoscopic Marking Using a New Marker, a Novel Luminomarker, in Lesion Marking Before Colorectal Cancer Surgery.
Acronym: Tattooing
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul St. Mary's Hospital (Other)
Collaborators: Hanlim Pharm. Co., Ltd. (Industry)
Responsible Party: Principal Investigator, In Kyeong Kim, Clinical Assistant Professor, Seoul St. Mary's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KC25MASI0456
Record Dates: First submitted 2025-12-21; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-12

CONDITIONS: Colorectal Cancer; Endoscopic Tattoo of Suspected Colon Cancer; Indocyanine Green (ICG)
Keywords: endoscopic tattooing; colorectal cancer; indocyanine green; LuminoMark
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: * Adult patients aged 19-80 years
  * Clinical T1-2, N0, without distant metastasis on imaging
  * If surgical treatment is required after ESD (endoscopic mucosal resection)*
  * If endoscopic lesion marking is required as determined by the attending physician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Luminomarker injection (Experimental): Through endoscopy, Luminomarker injection on submucosal layer. Location of injection : total 4 sites around tumor
  1. Left lateral side of tumor
  2. Right lateral side of tumor
  3. opposite of tumor (180 degree)
  4. distal part of 2cm from the tumor
  dosage of injection : at least 0.5cc per a site , total 2cc
  Interventions: Drug: LuminoMark inj. 0.2mL

INTERVENTIONS:
Drug: LuminoMark inj. 0.2mL — * Endoscopic tattooing with Luminomark on submucosal layer of bowel
  * Location of injection : total 4 sites
    1. Left lateral side of the tumor
    2. Right lateral side of the tumor
    3. opposite side of the tumor
    4. distal side of the tumor
  * Dosage of injection: -at least 0.5cc per a site, total 2ml

SUMMARY:
Early-stage lesions are difficult to identify intraoperatively during colorectal cancer surgery. Therefore, preoperative lesion marking using a colonoscopic approach is crucial to confirm the location and extent of resection during surgery. Preoperative lesion location can help determine the optimal extent of resection, thereby increasing the accuracy of colorectal surgery. This is particularly true for cases requiring surgery after early-stage colorectal cancer or endoscopic tumor resection. Therefore, preoperative marking with indocyanine green (IDG) allows for laparoscopic identification of the lesion. This is crucial because it allows for precise lesion location, thereby enhancing surgical accuracy and preventing the need for unnecessary additional resections.

DETAILED DESCRIPTION:
The recently developed indocyanine green (ICG)-hyaluronic acid mixture (LuminoMark™, Hanlim Pharm Co., Seoul, Republic of Korea) is a surgical marker combining indocyanine green with macroaggregated albumin (MAA). Its non-diffusing properties allow for precise lesion targeting. It addresses unmet needs of existing surgical markers, such as skin pigmentation and surgical site contamination. It effectively adsorbs onto cancerous lesions, enabling precise lesion location. Real-time tracking of the pigment allows for clear identification of the lesion's extent of removal, enhancing convenience and usability during surgery. It has already demonstrated superiority over existing labeling methods in a phase 3 clinical trial for breast lesions, receiving approval from the Ministry of Food and Drug Safety. Clinical trials are underway for various cancer types, including gastric and colon cancer, but it remains an over-approved drug.

Therefore, this study aimed to determine the accuracy of endoscopic labeling using a novel luminomarker for preoperative colon cancer lesion marking.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 19-80 years
* Clinical T1-2, N0, without distant metastasis on imaging
* If surgical treatment is required after ESD (endoscopic mucosal resection)*
* If endoscopic lesion marking is required as determined by the attending physician

Exclusion Criteria:

* Patients diagnosed with distant metastases (M1)
* Severe hepatic or renal dysfunction (Child-Pugh Class C, eGFR <39 mL/min/1.73 m2)
* Pregnant or lactating women
* High risk of intestinal obstruction or perforation
* Patients deemed inappropriate by the investigator (high-risk patients, such as patients with lung or heart disease, risk factors for bleeding, hepatitis virus infection, or other cancers)
* Patients with a history of hypersensitivity to the luminomarker drug or its components
* Patients who have experienced skin hypersensitivity to the dye
* Patients who do not wish to participate in the study

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-22 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Distance between endoscopic lesion markings and lesion location markings using luminomarkers for accuracy of tattooing | Perioperative/Periprocedural
  * Mix 1 vial (2 ml) of Indocyanine Green (ICG) + Hyaluronic Acid Mixture (Luminomarker™) with 1 vial (2 ml) of the attached solvent. Shake gently to dissolve thoroughly.
  * After performing an endoscopy to identify the lesion, attach the syringe to the endoscopic injector and mark at least three locations with at least 0.2 cc each.
  * After general anesthesia, insert a trocar for laparoscopic or robotic surgery and insert the laparoscopic equipment. Use a Laparoscopic near-intrared (NIR) camera to confirm the lesion marking.
  After marking with a surgical hemoclip, take a photograph and mark with a hemoclipping. A tumor is confirmed at the ICG-marked location in the obtained specimen.

SECONDARY OUTCOMES:
post-procedure related complication | through postoperative 4 days
  * Check for fever above 38°C (100°F) and abdominal pain before and after the procedure, and any abnormal findings such as free air on a simple X-ray.
  * Check for allergic reactions to medications.
  * Check for any postoperative complications and postoperative pathology results.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul St.Mary's hospital, the Catholic university of Korea, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided